CLINICAL TRIAL: NCT00351130
Title: An 8 Week Extension to a Randomized, Double-blind, Parallel Group, Active-controlled, Multi-center, 14 Week Study to Evaluate the Effectiveness of a Valsartan Versus and Amlodipine Treatment Strategy in Achieving Blood Pressure Control in Patients With Stage 1 or Stage 2 Hypertension or Uncontrolled on Present Monotherapy
Brief Title: Effectiveness of a Valsartan Based vs an Amlodipine Based Treatment Strategy in naïve Patients With Stage 1 or Stage 2 Hypertension or in Patients Uncontrolled on Current Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631B2406E1
Record Dates: First submitted 2006-03-16; First posted 2006-07-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension,; stage 1 hypertension,; stage 2 hypertension,; valsartan,; amlodipine,
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

INTERVENTIONS:
Drug: valsartan
Drug: amlodipine

SUMMARY:
Essential hypertension is a widespread disease which affects one out of every three adults in the industrialized world. It contributes to cardiovascular disease development, a major and well established risk factor. A patient non compliant to drug therapy is recognized as one of the primary reasons for inadequate blood pressure control.

ELIGIBILITY:
Inclusion criteria

* MSSBP> 140 mm Hg, and/or MSDBP> 90 mm Hg and currently treated with either valsartan 320 mg/ HCTZ 25 mg or amlodipine 10 mg/HCTZ 25 mg at end of core study

Exclusion criteria

* Premature discontinuation in the core study or failure to comply with the core study protocol
* Any patient that the investigator decides should not participate in the extension

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who reach BP goal, systolic <140 mmHg and diastolic <90 mmHg, after 22 weeks

SECONDARY OUTCOMES:
Percentage of patients who reach BP goal, systolic <140 mmHg and diastolic <90 mmHg, after 14 and 22 weeks
Adverse events after 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novatis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland